CLINICAL TRIAL: NCT00332618
Title: Multicenter Controlled Parallel-Groups Trial to Evaluate the Efficacy, Safety and Acceptability of TGO Buccal Spray Versus a Saliva Substitute in the Treatment of Psychotropic Medicines-Induced Xerostomia
Brief Title: Efficacy Study of Oxygenated Glycerol Triesters to Treat Xerostomia
Status: Completed | Type: Observational
Sponsor: Laboratoires CARILENE (Industry)
Other Study IDs: Laboratoires CARILENE
Record Dates: First submitted 2006-05-31; First posted 2006-06-01 (Estimated); Last update posted 2006-06-07 (Estimated); Status verified 2003-03

CONDITIONS: Xerostomia
Keywords: MULTICENTER; CONTROLLED; PARALLEL GROUPS
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Device: OXYGENATED GLYCEROL TRIESTERS

SUMMARY:
The objective of the trial was to evaluate the efficacy and clinical safety and acceptability of Oxygenated Glycerol Triesters in the relief of symptoms of xerostomia versus a reference comparator.

DETAILED DESCRIPTION:
Xerostomia is due to inadequate (hyposialia) or inexistent (asialia) saliva secretion.

There are may causes. Transitory xerostomia may occur in the presence of anxiety (stage fright, fear or dehydration). Prolonged xerostomia is most often related to a systemic disease, certain medicines or to radiotherapy of the head or neck.

Salivation depends upon the autonomic (sympathetic and parasympathetic) nervous system for its production and on the central nervous system for stimuli-dependant excretion. Substances acting on alpha an beta sympathetic receptors, whether agonists or antagonists, may induce hyposialia. Atropine, the main antagonist of the parasympathetic system, is present in many medicines used for pulmonary, ophthalmic or neurological purposes, potentially causing hyposialia. Similarly, imipramine antidepressants, phenothiazine neuroleptics, antihistamines and disopyramide predispose to the onset of hyposialia.

Xerostomia is often accompanied by buccal signs such as impaired sense of taste, halitosis and buccal ulcers and interferes with functions such as speech, chewing and swallowing. Because of reduced salivary secretion , there is a disturbance of the microbial colonization of the buccal cavity. Xerostomia has significant untoward effects on the buccal cavity and the quality of life of patients.

The basis of the treatment of xerostomia involves the use of saliva substitutes and/or saliva stimulants. Oxygenated Glycerol Triesters is neither a replacement for nor stimulant of saliva. It is a lubricant and protective solution for endobuccal spray.

ELIGIBILITY:
Inclusion Criteria:

* men or women over 18 years of age
* with a diagnosis requiring the prescription of psychotropies (antidepressants, tranquilizers, etc) for more than 6 weeks
* having received no palliative treatment for xerostomia for a minimum of the past 2 weeks
* having xerostomia meeting the questionnaire selection criteria and the sialometer method parameters
* patients legally competent to give their consent
* capable of and accepting to participate in the trial and capable of and accepting to answer trial questionnaires

Exclusion Criteria:

* combined treatments incompatible with the trial, un particular alcoholic solutions
* diabetes, any buccal condition requiring antimicrobial treatment
* Sjögren's syndrome or othermedical causes of xerostomia
* current participation in other clinical trials
* patient suffering from cancer
* patients with allergy to or known intolerance of any of the constituents of the investigational products
* patients treated with pilocarpine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74
Dates: Start 2003-09; Study Completion 2004-04

CONTACTS AND LOCATIONS:
Overall Officials: YVES YT TILLET, Expertpharma, Study Director — WHITE TILLET Consultants; Jean Baptiste JO Orler, Psychiatrist, Principal Investigator — CHU HOPITAL DES BROUSSAILLES
Locations (1):
- Chu Hopital Des Broussailles, Cannes, France

REFERENCES:
- [Background] Fox PC. Management of dry mouth. Dent Clin North Am. 1997 Oct;41(4):863-75. PMID 9344281